CLINICAL TRIAL: NCT06910904
Title: CONSTRAINT-INDUCED MOVEMENT THERAPY (CIMT) VS. MIRROR THERAPY (MT) ON HAND FUNCTION AND SPASTICITY IN PATIENTS WITH HEMIPARESIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lahore (Other)
Responsible Party: Principal Investigator, Mahnoor Aleem, Student, University of Lahore
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Rec-UOL-/495/08/24
Record Dates: First submitted 2025-03-28; First posted 2025-04-04 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-03

CONDITIONS: Stroke; Hemiparesis; Hemiparesis After Stroke
Keywords: Constraint-Induced Movement Therapy; Fugl-Meyer Assessment; Hemiparesis; Mirror Therapy; Spasticity
MeSH Terms: conditions — Stroke; Paresis; Muscle Spasticity | interventions — Constraint Induced Movement Therapy; Mirror Movement Therapy

STUDY DESIGN:
Intervention Model Description: This study employed a randomized, two-arm parallel interventional design to compare the effects of Constraint-Induced Movement Therapy (CIMT) and Mirror Therapy (MT) in patients with hemiparesis. Participants were randomly assigned to receive either CIMT or MT over an 8-week period, following standardized treatment protocols. Assessments were conducted at baseline, mid-point, and post-intervention using the Fugl-Meyer Assessment (FMA-UE) and Modified Ashworth Scale (MAS). The parallel group model ensured unbiased comparisons between the interventions, reflecting a practical clinical setting. This approach allowed for independent evaluation of each therapy's effectiveness on motor function and spasticity.
Who Masked: Outcomes Assessor
Masking Description: In this study, a single-blind design was implemented where the outcome assessors were masked to group allocation to reduce assessment bias. Participants and therapists delivering the interventions were not masked due to the nature of the therapies, which required active participation and visible techniques. Data analysts were also blinded to group identities during statistical processing to maintain objectivity. No additional parties beyond assessors and analysts were involved in masking.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Constraint-Induced Movement Therapy (CIMT) (Experimental): CIMT is a intensive training sessions of 6 hours/day for 5 weeks, focusing on functional tasks with the paretic arm while constraining the unaffected arm using a mitt or sling. Implement a constraint on the non-paretic arm to encourage increased use of the affected arm in daily activities.
  Interventions: Combination Product: Constraint-Induced Movement Therapy (CIMT)
- Mirror Therapy (MT) (Experimental): A specific intervention that uses a mirror to create a visual illusion of the affected limb, with the goal of improving motor function and quality of life in chronic stroke patients. In mirror therapy, the patient is asked to move the unaffected limb while watching the moving limb being reflected in the mirror.
  Interventions: Combination Product: Mirror Therapy (MT)

INTERVENTIONS:
Combination Product: Constraint-Induced Movement Therapy (CIMT) — CIMT is a intensive training sessions of 6 hours/day for 5 weeks, focusing on functional tasks with the paretic arm while constraining the unaffected arm using a mitt or sling. Implement a constraint on the non-paretic arm to encourage increased use of the affected arm in daily activities. Use shaping techniques to gradually increase the complexity and difficulty of tasks performed with the affected arm (Rahman, 2016). Most commonly, the protocol continues to be 2 weeks in duration but the intensity is adjusted such that the restraint is worn for approximately 6 h per day and therapy is administered for 2 to 3 h per day (MacKenzie & Viana, 2024). But this study implementing a 2 hour CIMT protocol with 6h restrain for 8 weeks in sub-acute stroke rehabilitation balances therapeutic intensity with practical considerations, potentially enhancing patient engagement and rehabilitation outcomes within clinical settings (Chen et al., 2014; Udoeyop, 2017).
  Arms: Constraint-Induced Movement Therapy (CIMT)
Combination Product: Mirror Therapy (MT) — A specific intervention that uses a mirror to create a visual illusion of the affected limb, with the goal of improving motor function and quality of life in chronic stroke patients. In mirror therapy, the patient is asked to move the unaffected limb while watching the moving limb being reflected in the mirror. The congruent visual feedback through the mirror affects brain lesions and motor-related areas on the affected side, facilitating motor recovery. Patients with chronic stroke who can benefit from visual feedback to enhance motor recovery (Gandhi et al., 2020; Rothgangel & Braun, 2013). Mirror therapy sessions should last at least 10 minutes daily, with the option to increase up to 30 minutes for optimal benefits. Practice mirror therapy exercises at least once a day. Perform gentle movements with the intact limb while observing its reflection in the mirror(Crosby et al., 2016).
  Arms: Mirror Therapy (MT)

SUMMARY:
This study aimed to compare the effects of Constraint-Induced Movement Therapy (CIMT) and Mirror Therapy (MT) on hand function and spasticity in individuals with hemiparesis. A total of 68 participants diagnosed with hemiparesis due to stroke or traumatic brain injury were recruited and randomly assigned to two equal groups. Group A received CIMT, while Group B underwent Mirror Therapy. Both interventions were administered over an 8-week period in a controlled rehabilitation setting. Functional assessments were conducted using the Fugl-Meyer Assessment for Upper Extremity (FMA-UE) to evaluate motor function and the Modified Ashworth Scale (MAS) to measure spasticity. Data collection occurred at baseline, the 4th week, and the 8th week of the intervention. Descriptive statistics were used to summarize demographic characteristics and baseline measurements, while inferential statistics, including repeated-measures ANOVA and independent t-tests, were applied to assess within- and between-group changes over time. The study also ensured assumptions of normality and sphericity were met to validate the statistical analyses. Demographic data such as age, gender, diagnosis type, and education level were also recorded to understand group comparability and potential influences on therapy outcomes. This study adds to the growing body of literature on non-invasive, evidence-based rehabilitation strategies for upper limb recovery.

DETAILED DESCRIPTION:
Hemiparesis, often resulting from conditions such as stroke or traumatic brain injury (TBI), leads to significant impairment in upper limb function and increased spasticity, adversely affecting daily living activities and overall quality of life. Rehabilitation strategies focusing on motor relearning, functional task training, and neuroplastic adaptation are crucial for regaining voluntary control and independence. Among the numerous interventions available, Constraint-Induced Movement Therapy (CIMT) and Mirror Therapy (MT) have emerged as two widely researched and clinically applied neurorehabilitation techniques targeting motor recovery in patients with hemiparesis.

Constraint-Induced Movement Therapy is based on the principle of "learned non-use," where the unaffected limb is restricted to encourage active use of the affected limb through repetitive, task-specific training. This therapy stimulates cortical reorganization and promotes motor recovery by intensively engaging the paretic limb. In contrast, Mirror Therapy involves the use of a mirror placed in the patient's midline to reflect movements of the unaffected limb, creating a visual illusion that the affected limb is functioning normally. This visual feedback mechanism is believed to activate mirror neurons and support motor relearning through sensory-motor integration.

This study was designed to compare the efficacy of CIMT and Mirror Therapy on improving hand function and reducing spasticity in patients with hemiparesis. The purpose was to determine whether one intervention offers superior functional outcomes or if both are equally beneficial, thereby informing evidence-based rehabilitation practices. A randomized, two-group design was employed to ensure balanced distribution and comparability between the intervention arms.

A total of 68 participants diagnosed with hemiparesis due to either ischemic stroke, hemorrhagic stroke, or traumatic brain injury were recruited from a rehabilitation center. Inclusion criteria involved patients aged 40-65 years with unilateral upper limb paresis, preserved cognitive function to follow instructions, and the ability to participate in scheduled therapy sessions. Exclusion criteria included individuals with severe cognitive deficits, unhealed fractures, or other orthopedic conditions that could interfere with upper limb training.

Participants were randomly allocated into two groups: Group A received Constraint-Induced Movement Therapy and Group B received Mirror Therapy. Both interventions were carried out over an 8-week period with standardized protocols. CIMT participants wore a mitt or sling on their unaffected limb for several hours each day during therapy to force usage of the affected arm in performing guided, functional tasks. Mirror Therapy participants performed symmetrical bilateral movements while focusing on the reflection of their unaffected arm in the mirror, tricking the brain into perceiving normal movement in the paretic limb.

Outcome measures were recorded at three time points: baseline (pre-intervention), 4th week (mid-intervention), and 8th week (post-intervention). The Fugl-Meyer Assessment for Upper Extremity (FMA-UE) was used to evaluate motor performance, coordination, and reflexes, serving as a standardized scale for upper limb motor recovery. To assess muscle tone and spasticity, the Modified Ashworth Scale (MAS) was employed. These validated tools allowed objective tracking of motor progress and spasticity changes throughout the intervention.

In addition to the primary outcome measures, the study collected comprehensive demographic and clinical data, including age, gender, diagnosis type, time since diagnosis, education level, employment status, and housing situation. These variables were recorded to assess baseline equivalence between groups and identify any confounding factors that might influence therapy outcomes.

Data were analyzed using SPSS software. Descriptive statistics were applied to summarize demographic characteristics and baseline data, including measures of central tendency and dispersion. Repeated-measures ANOVA was used to evaluate within-subject changes over time for each outcome measure, while independent t-tests assessed between-group differences at each time point. Tests for normality (Kolmogorov-Smirnov) and sphericity (Mauchly's Test) were performed to validate the assumptions for parametric analysis.

By directly comparing two commonly used interventions within the same clinical framework, this study sought to provide physiotherapists and clinicians with practical insights into selecting the most appropriate, evidence-based rehabilitation strategies for upper limb recovery in patients with hemiparesis. The structured design, standardized outcome measures, and comprehensive statistical analysis aimed to contribute meaningfully to the existing body of neurorehabilitation research.

ELIGIBILITY:
Inclusion Criteria:

* Participants having age (between 40 and 65 years old) will be recruited.
* Both gender were included (e Silva et al., 2017).
* Participants having ability to follow verbal and visual instructions (Danlami & Abdullahi, 2017).
* Patient having hemiparesis from 14 to 90 days (Bastola et al., 2021).
* Patients with mild to moderate spasticity (Burnstrom stage 2) (Jan et al., 2019).
* Patients experiencing functional limitations in hand motor function (Gracies et al., 2019).

Exclusion Criteria:

* History of other neurological conditions (Mansfield et al., 2018).
* Unstable fracture or other orthopedic conditions (Page et al., 2007).
* Individuals with physical limitations that prevent them from positioning themselves adequately to view their affected limb in the mirror during therapy sessions, as this could compromise the effectiveness of mirror therapy (Danlami & Abdullahi, 2017).
* History of shoulder instability or major orthopedic surgery in the affected arm (Gracies et al., 2019).

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2024-09-15 (Actual); Primary Completion 2025-03-19 (Actual); Study Completion 2025-03-28 (Actual)

PRIMARY OUTCOMES:
Motor impairment and and joint functioning | Baseline, Week 4, and Week 8
  Assessed using the Fugl-Meyer Assessment for Upper Extremity (FMA-UE), which measures motor function, coordination, and reflex activity in the affected limb to evaluate improvements in voluntary movement.

SECONDARY OUTCOMES:
Spasticity | Baseline, Week 4, and Week 8
  Measured using the Modified Ashworth Scale (MAS), which assesses muscle tone and resistance during passive soft-tissue stretching. It evaluates changes in spasticity levels of the affected upper limb over time.

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Lahore Teaching Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Chen YP, Pope S, Tyler D, Warren GL. Effectiveness of constraint-induced movement therapy on upper-extremity function in children with cerebral palsy: a systematic review and meta-analysis of randomized controlled trials. Clin Rehabil. 2014 Oct;28(10):939-53. doi: 10.1177/0269215514544982. Epub 2014 Aug 14. PMID 25125440